CLINICAL TRIAL: NCT00382408
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Efficacy, and Immunogenicity of DR-5001
Brief Title: A Clinical Trial to Evaluate the Safety, Efficacy, and Immunogenicity of DR-5001
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DR-ADV-301
Record Dates: First submitted 2006-09-27; First posted 2006-09-29 (Estimated); Results first posted 2012-05-25 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-03

CONDITIONS: Respiratory Tract Diseases
Keywords: Acute respiratory disease prevention; Adenovirus
MeSH Terms: conditions — Respiratory Tract Diseases; Adenoviridae Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccine (Experimental): Participants received a single tablet of both Type-4 and Type-7 adenovirus vaccines at study visit 1 (Day 0).
  Interventions: Biological: DR-5001
- Placebo (Placebo Comparator): Participants received a single tablet of both placebos that matched the Type-4 and Type-7 adenovirus vaccines at study visit 1 (Day 0).
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: DR-5001 — All randomized subjects received a single tablet of both Type-4 and Type-7 ADV vaccines on Day 0. Both vaccine tablets were administered orally, kept in the mouth as briefly as possible and swallowed whole with water. Chewing the tablets was not permitted.
  Arms: Vaccine
Other: Placebo — All randomized subjects received a single tablet each of the placebos matching Type-4 and Type-7 ADV vaccines on Day 0. Both placebo tablets were administered orally, kept in the mouth as briefly as possible and swallowed whole with water. Chewing the tablets was not permitted.
  Arms: Placebo

SUMMARY:
This is a multicenter, double-blind, randomized, placebo-controlled study to evaluate the safety and efficacy of oral DR-5001 in reducing the attack rate of febrile acute respiratory disease caused by type-4 and type-7 adenovirus as well as determine its immunogenicity.

DETAILED DESCRIPTION:
The study will be conducted at two sites and will include a minimum of 4 visits. The overall study duration for participants will be approximately 8 weeks. Study participants will undergo acute respiratory disease evaluation that will include a throat swab and a blood draw. Each participant will also be contacted in six months for follow-up information.

ELIGIBILITY:
Inclusion Criteria:

* Military recruit in training
* Male or female; if female, must be of non-childbearing potential or with a documented negative pregnancy test </= 72 hours prior to study medication administration and agree not to become pregnant

Exclusion Criteria:

* Female nursing an infant or planning on nursing during the study
* Immunosuppressed for any reason, including past (within last 6 months) or current treatment with immunosuppressive therapy
* Known allergy to any component of the vaccines and/or placebo tablets
* Immunocompromised sexual partner or immunocompromised individuals in home

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4040 (Actual)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duramed Protocol Chair, Study Chair — Duramed Research, Inc.
Locations (2):
- United States (2):
  - Duramed Investigational Site, Great Lakes, Illinois
  - Duramed Investigational Site, Fort Jackson, South Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in subjects undergoing military basic training.
Pre-assignment Details: Participants were randomized to either the vaccine group or the matching placebo group in a 3:1 ratio.
Period: Overall Study
Arm/Group | Vaccine | Placebo
Started | 3031 | 1009
Completed | 2887 | 955
Not Completed | 144 | 54
Not completed — Did not meet protocol requirement | 3 | 3
Not completed — Protocol Violation | 2 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 17 | 6
Not completed — Pregnancy | 2 | 0
Not completed — Lost to Follow-up | 19 | 8
Not completed — Other | 100 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccine | Placebo | Total
Number analyzed (Participants) | 3031 | 1009 | 4040
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.3 (4.0) | 21.1 (4.1) | 21.2 (4.0)
Age, Customized [Median (Full Range); unit: years] | 19.8 [17.1 to 42.0] | 19.7 [17.1 to 42.2] | 19.8 [17.1 to 42.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1121 | 367 | 1488
  Male | 1910 | 642 | 2552
Race/Ethnicity, Customized [Number; unit: participants]
  African-American | 554 | 186 | 740
  Asian | 94 | 29 | 123
  Caucasian | 1871 | 642 | 2513
  Hispanic | 326 | 103 | 429
  Other | 186 | 49 | 235
Region of Enrollment [Number; unit: participants]
  United States | 3031 | 1009 | 4040
Type-4 Titer [Number; unit: participants] — Negative = titer value <1:4 Positive = titer value >=1:4
  participants
    Negative | 1906 | 678 | 2584
    Positive | 1123 | 331 | 1454
    Unknown | 2 | 0 | 2
Type-7 Titer [Number; unit: participants] — Negative = titer value <1:4 Positive = titer value >=1:4
  participants
    Negative | 1159 | 377 | 1536
    Positive | 1870 | 632 | 2502
    Unknown | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Wild Type-4 Febrile Adenovirus (ADV) Acute Respiratory Disease (ARD) -- ITT Cohort
Description: For the oral Type-4 vaccine, the primary outcome is the number of cases of ADV-4 febrile acute respiratory disease (ARD), defined as a subject with one or more clinical signs and symptoms of ARD and an oral temperature ≥ 100.5°F (38.06°C) and throat culture positive for wild ADV Type-4 infection. This outcome used the intent-to-treat cohort.
Time Frame: Day 0 - Day 56
Population: The intent-to-treat (ITT) cohort included all participants randomized and treated in the study.
Measure: Number; unit: participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 3031 | 1009
participants | 1 | 48
Statistical Analysis 1: Comparison: Vaccine vs Placebo; The vaccine efficacy (VE) was defined as: VE = 1 - R, where R = P(vaccine)/P(placebo) was the relative risk of ARD attack in subjects who received vaccines compared to placebos (Blackwelder 1993). The 95% confidence interval of the VE was obtained by inverting the Chi Square method proposed by Koopman for the ratio of two binomial proportions (Koopman 1984). The goal of the analysis of efficacy was to demonstrate a VE of at least 80% with a lower 95% confidence bound at least 60%; Test type: Superiority or Other; vaccine efficacy (VE) = 99.31, 95% CI 2-sided [96.02 to 99.88]

2. Primary Outcome: Number of Participants With Wild Type-4 Febrile Adenovirus (ADV) Acute Respiratory Disease (ARD) -- PP Cohort
Description: For the oral Type-4 vaccine, the primary outcome is the number of cases of ADV-4 febrile acute respiratory disease (ARD), defined as a subject with one or more clinical signs and symptoms of ARD and an oral temperature ≥ 100.5°F (38.06°C) and throat culture positive for wild ADV Type-4 infection. This outcome used the per protocol cohort.
Time Frame: Day 0 - Day 56
Population: The per-protocol (PP) cohort included all participants who met the eligibility criteria set forth in the protocol, did not have any significant violations or deviations from the protocol, and completed the final study visit (Day 56). Subjects who vomited within 24 hours after taking the study medication were excluded from the PP cohort.
Measure: Number; unit: participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 2855 | 945
participants | 1 | 47

3. Primary Outcome: Number of Participants With Wild Type-4 Febrile Adenovirus (ADV) Acute Respiratory Disease (ARD) -- ITT Cohort --- Day 11-56
Description: For the oral Type-4 vaccine, the primary outcome is the number of cases of ADV-4 febrile acute respiratory disease (ARD), defined as a subject with one or more clinical signs and symptoms of ARD and an oral temperature ≥ 100.5°F (38.06°C) and throat culture positive for wild ADV Type-4 infection. This outcome used the intent-to-treat cohort; further, this outcome omitted ARD cases from Day 0-Day 10 because the protective effect of the vaccine was unlikely to take place during that time period.
Time Frame: Day 11 - Day 56
Population: The intent-to-treat (ITT) cohort included all participants randomized and treated in the study.
Measure: Number; unit: participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 3031 | 1009
participants | 0 | 44

4. Primary Outcome: Percentage of Participants Showing ADV-7 Seroconversion at Week 4
Description: ADV-7 seroconversion was defined as the development of ADV Type-7 neutralizing antibody at Week 4 (Day 26) after study medication that represented at least a fourfold increase in titer from baseline (visit 0) in a subject whose baseline Type-7 titer was <1:4.
Time Frame: Week 4
Population: Type-7 ADV Seroconversion Cohort: Included those subjects who had a negative Type-7 ADV serum neutralizing antibody status at baseline (<1:4) and at least one titer value for ADV-7 at the subsequent visits following vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 1120 | 359
percentage of participants | 93.8 [92.4 to 95.2] | 5.3 [3.0 to 7.6]

5. Secondary Outcome: Percentage of Participants Showing ADV-4 Seroconversion at Week 4
Description: ADV-4 seroconversion was defined as the development of ADV Type-4 neutralizing antibody at Week 4 (Day 26) after study medication that represented at least a fourfold increase in titer from baseline (visit 0) in a subject whose baseline Type-4 titer was <1:4.
Time Frame: Week 4
Population: Type-4 ADV Seroconversion Cohort: Included those subjects who had a negative Type-4 ADV serum neutralizing antibody status at baseline (<1:4) and at least one titer value for ADV-4 at the subsequent visits following vaccination.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 1841 | 653
percentage of participants | 94.5 [93.4 to 95.5] | 10.6 [8.2 to 12.9]

6. Secondary Outcome: Number of Participants With Wild Type-4 Adenovirus (ADV) Acute Respiratory Disease (ARD) -- ITT Cohort
Description: For the oral Type-4 vaccine, the number of cases of ADV-4 acute respiratory disease (ARD) regardless of whether the participant was febrile or not. Therefore includes participants with one or more clinical signs and symptoms of ARD and throat culture positive for wild ADV Type-4 infection. This outcome used the intent-to-treat cohort.
Time Frame: Day 0 - Day 56
Population: The intent-to-treat (ITT) cohort included all participants randomized and treated in the study.
Measure: Number; unit: participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 3031 | 1009
participants | 3 | 65
Statistical Analysis 1: Comparison: Vaccine vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; vaccine efficacy (VE) = 98.46, 95% CI 2-sided [95.39 to 99.49]

7. Secondary Outcome: Percentage of Participants Showing ADV Type-4 Booster at Week 4
Description: ADV-4 booster effect is defined as the development of ADV Type-4 neutralizing antibody at Week 4 (Day 26) that represented at least a fourfold increase in titer from baseline (Visit 0) in a participant whose baseline Type-4 titer is ≥1:4.
Time Frame: Baseline, Week 4
Population: Type-4 ADV Booster Cohort included subjects who had a positive Type-4 ADV serum neutralizing antibody status at baseline (≥ 1:4) and at least one titer value for ADV Type-4 at the subsequent visits following study medication administration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 1094 | 326
percentage of participants | 50.3 [47.3 to 53.2] | 0.6 [-0.2 to 1.5]

8. Secondary Outcome: Number of Participants With Wild Type-7 Febrile Adenovirus (ADV) Acute Respiratory Disease (ARD) -- ITT Cohort
Description: For the oral Type-7 vaccine, a secondary outcome is the number of cases of ADV-7 febrile acute respiratory disease (ARD), defined as a subject with one or more clinical signs and symptoms of ARD and an oral temperature ≥ 100.5°F (38.06°C) and throat culture positive for wild ADV Type-7 infection. This outcome used the intent-to-treat cohort.
Time Frame: Day 0 - Day 56
Population: The intent-to-treat (ITT) cohort included all participants randomized and treated in the study.
Measure: Number; unit: participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 3031 | 1009
participants | 0 | 0

9. Secondary Outcome: Number of Participants With Wild Type-7 Adenovirus (ADV) Acute Respiratory Disease (ARD) -- ITT Cohort
Description: For the oral Type-7 vaccine, the number of cases of ADV-7 acute respiratory disease (ARD) regardless of whether the participant was febrile or not. Therefore includes participants with one or more clinical signs and symptoms of ARD and throat culture positive for wild ADV Type-7 infection. This outcome used the intent-to-treat cohort.
Time Frame: Day 0 - Day 56
Population: The intent-to-treat (ITT) cohort included all participants randomized and treated in the study.
Measure: Number; unit: participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 3031 | 1009
participants | 0 | 0

10. Secondary Outcome: Percentage of Participants Showing ADV Type-7 Booster at Week 4
Description: ADV-7 booster effect is defined as the development of ADV Type-7 neutralizing antibody at Week 4 (Day 26) that represented at least a fourfold increase in titer from baseline (Visit 0) in a participant whose baseline Type-7 titer is ≥1:4.
Time Frame: Baseline, Week 4
Population: Type-7 ADV Booster Cohort included subjects who had a positive Type-7 ADV serum neutralizing antibody status at baseline (≥ 1:4) and at least one titer value for ADV Type-7 at the subsequent visits following study medication administration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 1815 | 620
percentage of participants | 46.1 [43.8 to 48.4] | 3.9 [2.4 to 5.4]

ADVERSE EVENTS:
Time Frame: Day 0 (vaccination day) - Day 56
Arm/Group | Placebo | Vaccine
Serious Adverse Events (participants affected / at risk) | 12/1009 | 35/3031
Other Adverse Events (participants affected / at risk) | 916/1009 | 2673/3031
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=1009) | Vaccine (N=3031)
BASEDOW'S DISEASE (Endocrine disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (2)
HERNIA (General disorders) | 0 (0) | 1 (1)
FOOD ALLERGY (Immune system disorders) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 1 (1) | 1 (1)
BRONCHITIS ACUTE (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1) | 2 (2)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 2 (2)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 1 (1)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1 (1) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CONCUSSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
JAW FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
LIGAMENT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
STRUCK BY LIGHTNING (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ADJUSTMENT DISORDER (Psychiatric disorders) | 0 (0) | 3 (3)
ADJUSTMENT DISORDER WITH ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0)
ADJUSTMENT DISORDER WITH DEPRESSED MOOD (Psychiatric disorders) | 0 (0) | 1 (1)
ADJUSTMENT DISORDER WITH MIXED ANXIETY AND DEPRESSED MOOD (Psychiatric disorders) | 0 (0) | 1 (1)
BIPOLAR DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
CYCLOTHYMIC DISORDER (Psychiatric disorders) | 0 (0) | 1 (1)
DEPRESSED MOOD (Psychiatric disorders) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1)
MAJOR DEPRESSION (Psychiatric disorders) | 1 (1) | 1 (1)
PERSONALITY DISORDER (Psychiatric disorders) | 0 (0) | 1 (1)
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
STRESS (Psychiatric disorders) | 1 (1) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 1 (1)
SUICIDE ATTEMPT (Psychiatric disorders) | 2 (2) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=1009) | Vaccine (N=3031)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 175 (216) | 482 (593)
DIARRHOEA (Gastrointestinal disorders) | 112 (142) | 387 (484)
NAUSEA (Gastrointestinal disorders) | 193 (246) | 552 (654)
VOMITING (Gastrointestinal disorders) | 68 (77) | 181 (209)
CHILLS (General disorders) | 55 (56) | 84 (86)
PYREXIA (General disorders) | 60 (60) | 139 (146)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 424 (490) | 1193 (1361)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 131 (134) | 475 (493)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 270 (372) | 787 (1070)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 55 (57) | 110 (113)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 72 (79) | 233 (254)
HEADACHE (Nervous system disorders) | 447 (659) | 1237 (1795)
COUGH (Respiratory, thoracic and mediastinal disorders) | 238 (294) | 685 (855)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 226 (273) | 740 (927)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 233 (271) | 743 (912)

LIMITATIONS AND CAVEATS:
In the past 6 years, Type-7 ADV has only rarely been recovered from recruits with ARD (Russell 2007). Therefore, it may not be possible to directly measure the protective effect of the vaccine against Type-7 ADV in the proposed study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can (i) review results communications prior to public release and can embargo communications regarding trial results for a period of at least 60 days but no more than 180 days from the time submitted to the sponsor for review; and (ii) require in instances of a multi-center study, that a single PI not disclose study data until after the multi-center results are published, provided such results are published within eighteen (18) months of the conclusion of the study.